CLINICAL TRIAL: NCT07335185
Title: Gravity Stroke System for Recanalization of Large Vessel Occlusion Strokes
Acronym: GRASSROOT Reg
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gravity Medical Technology, INC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMT-GRASSROOT-2026-01
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Ischemic Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Disease
Keywords: Mechanical Thrombectomy; Brain; Brain Clot; Cerebral Ischemia; Brain Infarction; Neurovascular Intervention; Revascularization; Reperfusion; Stent Retriever; Supernova; Stroke; Gravity Medical Technology
MeSH Terms: conditions — Stroke; Ischemic Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Brain Ischemia; Brain Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supernova revascularization device (Experimental): Mechanical thrombectomy with Supernova Stent Retriever
  Interventions: Device: Supernova revascularization device

INTERVENTIONS:
Device: Supernova revascularization device — Mechanical Thrombectomy

SUMMARY:
Supernova and Neutron are endovascular mechanical revascularization devices indicated to restore blood flow by removing thrombus from a large intracranial vessel in patients experiencing an acute ischemic stroke within 24 hours of symptom onset or from last known well time.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has experienced an Acute Ischemic Stroke due to large intracranial vessel occlusion in at least one of the following intracranial vessels: internal carotid artery (ICA), M1and M2 segments of the middle cerebral artery (MCA), basilar, and vertebral artery.
2. Subject has been or will be treated with Supernova and/or Neutron devices as the initial device used to remove the thrombus
3. Subject is willing to participate in a 90-day follow-up visit.

Exclusion Criteria:

* Concurrent participation in another mechanical neurothrombectomy device trial or any other clinical trial with an active treatment arm where the study procedure or treatment might confound the results of the registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-10-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful reperfusion | Day 0 (end of procedure)
  Rate of successful reperfusion, defined as modified Thrombolysis in Cerebral Ischemia (mTICI) grade of 2b or higher
  Grade 0: No reperfusion Grade 3: Complete reperfusion
Symptomatic intracranial hemorrhage | sICH measured within 24 (18-36) hours of the procedure
  Safety (Rate of symptomatic intracranial hemorrhage (sICH) as measured by the SITS-MOST criteria) The SITS-MOST definition of SICH is a local or remote type II parenchymal haemorrhage within 22 to 36 hours after treatment (or sooner) associated with a ≥ fourpoint deterioration on the NIHSS score from baseline or from the lowest score from baseline to 24 hours, or leading to death.
All-cause mortality | All-cause mortality measured at 90 (±14) days
  Safety (All-cause mortality)

SECONDARY OUTCOMES:
Percentage of participants with a modified Rankin Scale (mRS) score of ≤2 | 90 (±14) days post-treatment
  Effectiveness
  (The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death.
  Score 0: No symptoms Score 1: No significant disability. Able to carry out all usual activities, despite some symptoms.
  Score 2: Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  Score 3: Moderate disability. Requires some help, but able to walk unassisted. Score 4: Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  Score 5: Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  Score 6: Dead)
Asymptomatic Intracranial Hemorrhage | Day 1 (within 24 hours (18-36 hours) of the procedure)
  Incidence of any asymptomatic intracranial hemorrhage post-procedure
Neurological Deterioration | Day 1 (within 24 hours (18-36 hours) of the procedure)
  Safety (defined as a ≥4-point increase in the National Institutes of Health Stroke Scale (NIHSS) score)

IPD SHARING:
Plan to Share IPD: No